CLINICAL TRIAL: NCT00881361
Title: A Phase II Study Evaluating the Role of Sentinel Lymph Node Surgery and Axillary Lymph Node Dissection Following Preoperative Chemotherapy in Women With Node Positive Breast Cancer (T1-4, N1-2, M0) at Initial Diagnosis
Brief Title: Surgery to Remove the Sentinel Lymph Node and Axillary Lymph Nodes After Chemotherapy in Treating Women With Stage II, Stage IIIA, or Stage IIIB Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOSOG-Z1071; ACOSOG-Z1071; CDR0000640100 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Sentinel Lymph Node Biopsy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study cohort (Other): Patients who plan to receive or have received neoadjuvant chemotherapy are eligible. Patients undergo examination for breast and axilla lymph adenopathy and then undergo ultrasound of the axillary nodes at baseline and after completion of neoadjuvant chemotherapy. Within 12 weeks of completing neoadjuvant chemotherapy, patients undergo a mastectomy or lumpectomy (per surgeon discretion) including both sentinel lymph node surgery and axillary lymph node dissection.
  Interventions: Drug: systemic chemotherapy; Procedure: axillary lymph node dissection; Procedure: neoadjuvant therapy; Procedure: sentinel lymph node biopsy; Procedure: therapeutic conventional surgery; Procedure: ultrasound imaging

INTERVENTIONS:
Drug: systemic chemotherapy
Procedure: axillary lymph node dissection
Procedure: neoadjuvant therapy
Procedure: sentinel lymph node biopsy
Procedure: therapeutic conventional surgery
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying surgery to remove the sentinel lymph node and axillary lymph nodes after chemotherapy in treating women with stage II, stage IIIA, or stage IIIB breast cancer.

DETAILED DESCRIPTION:
This is a multicenter study. Patients who plan to receive or have received neoadjuvant chemotherapy are eligible. Patients undergo examination for breast and axilla lymph adenopathy and then undergo ultrasound of the axillary nodes prior to registration to confirm eligibility and after completion of neoadjuvant chemotherapy. Within 12 weeks of completing neoadjuvant chemotherapy, patients undergo a mastectomy or lumpectomy (per surgeon discretion) including both sentinel lymph node surgery and axillary lymph node dissection. The primary and secondary objectives of the study are described below.

Primary Objective:

1. To determine the false negative rate for sentinel lymph node (SLN) surgery. Among the patients who have at least one sentinel lymph node identified and removed, false negative rate is defined as the number of patients declared to have no evidence of cancer in the SLN and are found to have at least one positive lymph node in the ALND divided by the total number of patients with at least one positive axillary lymph node by ALND.

Secondary Objectives:

1. To determine how the axillary ultrasound status of the patient upon completion of preoperative chemotherapy (evidence of residual lymphadenopathy on the ultrasound examination versus no evidence of lymphadenopathy in the ultrasound examination) affects the false negative rate of SLN and how sonographic findings correlate with residual disease on final pathology.
2. To determine the node status of patients after preoperative chemotherapy. Patients will be classified as node positive if they were determined to have at least one positive lymph node by SLN or ALND. Patients will be classified as node negative if all nodes examined by SLN and ALND were negative.
3. To determine whether the false-negative rate for SLN surgery after preoperative chemotherapy is related to the extent of residual cancer burden (RCB) overall, or separately in the breast or regional nodal basin.
4. To evaluate pathological complete response (pCR) rates (defined as no invasive disease in breast or lymph nodes) and disease-free survival (DFS) rates in node-positive patients receiving preoperative chemotherapy.

After completion of surgery, patients will visit the office for follow-up exams at 1-2 weeks then patients are followed every 6 months for 2 years, yearly for 2 years, then every other year for 6 years. The study closed to accrual and treatment on 5/29/12.

ELIGIBILITY:
Eligibility Criteria:

1. ≥ 18 years old
2. ECOG/Zubrod Performance Status 0-1
3. Female. Note: Men are excluded from this study because the number of men with breast cancer is insufficient to provide a statistical basis for assessment of effects in this subpopulation of people with breast cancer.
4. Histologic diagnosis of invasive breast cancer, clinical stage T0-4 N1-2 M0 (excluding inflammatory breast cancer).
5. FNA biopsy or core needle biopsy of an axillary node documenting nodal disease at time of diagnosis and prior to preoperative chemotherapy.
6. Preoperative chemotherapy must be completed or planned for patient. NOTE: Patients enrolling on studies involving preoperative chemotherapy (through cooperative groups or institutional studies) may be eligible for this study, provided sentinel node surgery prior to preoperative chemotherapy was not required in the other studies.
7. No prior ipsilateral axillary surgery, such as excisional biopsy of lymph node(s) or treatment of hidradenitis.
8. No prior SLN surgery/excisional lymph node biopsy for pathological confirmation of axillary status.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Boughey, MD, Study Chair — Mayo Clinic
Locations (324):
- United States (324):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Valley Medical Oncology, Fremont, California
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Community Hospital of the Monterey Peninsula Comprehensive Cancer Center, Monterey, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Sharp Memorial Hospital Cancer Center, San Diego, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Stanford Cancer Center, Stanford, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Robert and Carol Weissman Cancer Center at Martin Memorial, Stuart, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Clarian West Medical Center, Avon, Indiana
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Clarian North Medical Center, Carmel, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Maine Medical Center - Bramhall Campus, Portland, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Dyson Center for Cancer Care at Vassar Brothers Medical Center, Poughkeepsie, New York
  - Saint Francis Hospital Cancer Center, Poughkeepsie, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital Cancer Treatment Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Hilton Head Regional Medical Center, Hilton Head Island, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Nashville Breast Center, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Baptist Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Surgical Oncology Associates, Newport News, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Aurora Women's Pavilion of West Allis Memorial Hospital, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

REFERENCES:
- [Result] Le-Petross HT, McCall LM, Hunt K, et al.: Role of axillary ultrasound after neoadjuvant chemotherapy in women with node-positive breast cancer (T1-4, N1-2, M0) at initial diagnosis (ACOSOG Z1071). [Abstract] J Clin Oncol 30 (Suppl 15): A-1107, 2012.
- [Result] Boughey JC, Suman VJ, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Kuerer HM, Bowling M, Flippo-Morton TS, Byrd DR, Ollila DW, Julian TB, McLaughlin SA, McCall L, Symmans WF, Le-Petross HT, Haffty BG, Buchholz TA, Nelson H, Hunt KK; Alliance for Clinical Trials in Oncology. Sentinel lymph node surgery after neoadjuvant chemotherapy in patients with node-positive breast cancer: the ACOSOG Z1071 (Alliance) clinical trial. JAMA. 2013 Oct 9;310(14):1455-61. doi: 10.1001/jama.2013.278932. PMID 24101169
- [Result] Boughey JC, Ballman KV, Hunt KK, McCall LM, Mittendorf EA, Ahrendt GM, Wilke LG, Le-Petross HT. Axillary Ultrasound After Neoadjuvant Chemotherapy and Its Impact on Sentinel Lymph Node Surgery: Results From the American College of Surgeons Oncology Group Z1071 Trial (Alliance). J Clin Oncol. 2015 Oct 20;33(30):3386-93. doi: 10.1200/JCO.2014.57.8401. Epub 2015 Feb 2. PMID 25646192
- [Derived] Armer JM, Ballman KV, McCall L, Armer NC, Sun Y, Udmuangpia T, Hunt KK, Mittendorf EA, Byrd DR, Julian TB, Boughey JC. Lymphedema symptoms and limb measurement changes in breast cancer survivors treated with neoadjuvant chemotherapy and axillary dissection: results of American College of Surgeons Oncology Group (ACOSOG) Z1071 (Alliance) substudy. Support Care Cancer. 2019 Feb;27(2):495-503. doi: 10.1007/s00520-018-4334-7. Epub 2018 Jul 6. PMID 29980907
- [Derived] Boughey JC, Ballman KV, McCall LM, Mittendorf EA, Symmans WF, Julian TB, Byrd D, Hunt KK. Tumor Biology and Response to Chemotherapy Impact Breast Cancer-specific Survival in Node-positive Breast Cancer Patients Treated With Neoadjuvant Chemotherapy: Long-term Follow-up From ACOSOG Z1071 (Alliance). Ann Surg. 2017 Oct;266(4):667-676. doi: 10.1097/SLA.0000000000002373. PMID 28657941
- [Derived] Boughey JC, Suman VJ, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Flippo-Morton TS, Kuerer HM, Bowling M, Hunt KK; Alliance for Clinical Trials in Oncology. Factors affecting sentinel lymph node identification rate after neoadjuvant chemotherapy for breast cancer patients enrolled in ACOSOG Z1071 (Alliance). Ann Surg. 2015 Mar;261(3):547-52. doi: 10.1097/SLA.0000000000000551. PMID 25664534

RESULTS

PARTICIPANT FLOW:
Groups:
- cN1 Cohort: Patients who were staged according to the AJCC staging system as cN1 (disease in movable axillary lymph nodes) and plan to receive or have received neoadjuvant chemotherapy are eligible. Patients undergo examination for breast and axilla lymph adenopathy and then undergo ultrasound of the axillary nodes at baseline and after completion of neoadjuvant chemotherapy. Within 12 weeks of completing neoadjuvant chemotherapy, patients undergo a mastectomy or lumpectomy (per surgeon discretion) including both sentinel lymph node surgery and axillary lymph node dissection.
- cN2 Cohort: Patients who were staged according to the AJCC staging system as cN2 (disease in fixed or matted axillary lymph nodes) and plan to receive or have received neoadjuvant chemotherapy are eligible. Patients undergo examination for breast and axilla lymph adenopathy and then undergo ultrasound of the axillary nodes at baseline and after completion of neoadjuvant chemotherapy. Within 12 weeks of completing neoadjuvant chemotherapy, patients undergo a mastectomy or lumpectomy (per surgeon discretion) including both sentinel lymph node surgery and axillary lymph node dissection.
- cN3 Patients (Ineligible): Patients who were staged according to the AJCC staging system as cN3.
Period: Overall Study
Arm/Group | cN1 Cohort | cN2 Cohort | cN3 Patients (Ineligible)
Started | 707 | 47 | 2
Completed | 663 | 38 | 0
Not Completed | 44 | 9 | 2
Not completed — Terminated prior to surgery | 27 | 7 | 0
Not completed — Ineligible | 17 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Only cN1 and cN2 patients who completed the study were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | cN1 Cohort | cN2 Cohort | Total
Number analyzed (Participants) | 663 | 38 | 701
Age, Customized [Number; unit: participants]
  18-39 years old | 120 | 4 | 124
  40-49 years old | 213 | 15 | 228
  50-59 years old | 197 | 10 | 207
  60-69 years old | 112 | 5 | 117
  greater than 70 years old | 21 | 4 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 663 | 38 | 701
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 663 | 38 | 701

OUTCOME MEASURES:

1. Primary Outcome: False Negative Rate (FNR) for Sentinel Lymph Node (SLN) Surgery After Chemotherapy When at Least 2 SLNs Were Excised in Women Initially Presenting With Biopsy-proven cN1 Breast Cancer [cN1 Cohort]
Description: False negative rate (FNR) (percentage) for sentinel lymph node (SLN) surgery after chemotherapy when at least 2 SLNs were excised in women initially presenting with biopsy-proven cN1 breast cancer, defined as the number of patients with no positive lymph nodes by SLN and with at least one positive lymph node by axillary lymph node dissection (ALND) divided by the total number of patients initially presenting with biopsy-proven cN1 breast cancer with at least one positive lymph node by SLN or ALND multiplied by 100. A 2-sided Bayesian credible interval (BCI) for the true FNR was constructed.
Time Frame: At time of surgery
Population: Of the cN1 Cohort patients who Started the study (see Participant Flow), only patients with residual nodal disease were included in this analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | cN1 Cohort
Number analyzed (Participants) | 525
percentage of participants | 12.6 [9.85 to 16.05]

2. Secondary Outcome: False Negative Rate (FNR) for Sentinel Lymph Node (SLN) Surgery After Chemotherapy When at Least 2 SLNs Were Excised in Women Initially Presenting With Biopsy-proven cN2 Breast Cancer [cN2 Cohort]
Description: False negative rate (FNR) (percentage) for sentinel lymph node (SLN) surgery after chemotherapy when at least 2 SLNs were excised in women initially presenting with biopsy-proven cN2 breast cancer, defined as the number of patients with no positive lymph nodes by SLN and with at least one positive lymph node by axillary lymph node dissection (ALND) divided by the total number of patients initially presenting with biopsy-proven cN1 breast cancer with at least one positive lymph node by SLN or ALND multiplied by 100. An interval estimate of the SLN false negative rate will be constructed using the Duffy-Santner approach.
Time Frame: At time of surgery
Population: Of the cN2 Cohort patients who Started the study (see Participant Flow), only patients with residual nodal disease were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of false-negative SLN finding
Arm/Group | cN2 Cohort
Number analyzed (Participants) | 38
percentage of false-negative SLN finding | 0 [0 to 23.2]

3. Secondary Outcome: False-negative Rate (FNR) Under the Selection Process by Axillary Ultrasound (AUS) Status After Completion of Neoadjuvant Chemotherapy (NAC)
Description: False negative rate (FNR) (percentage) for sentinel lymph node (SLN) surgery after chemotherapy in women with normal AUS and at least 2 SLNs were excised, defined as the number of patients with no positive lymph nodes by SLN and with at least one positive lymph node by axillary lymph node dissection (ALND) divided by the total number of patients with at least one positive lymph node by SLN or ALND multiplied by 100.
Time Frame: At the time of surgery
Measure: Number (90% Confidence Interval); unit: percentage of false-negative SLN finding
Groups:
- Post-chemotherapy AUS Normal: Patients with lymph nodes classified as normal if the radiologist was unable to visualize any lymph nodes on axillary ultrasound (AUS) or indicated that the lymph nodes were normal in morphologic appearance.
Arm/Group | Post-chemotherapy AUS Normal
Number analyzed (Participants) | 470
percentage of false-negative SLN finding | 12.6 [9.5 to 16.3]

4. Secondary Outcome: Node Status After Preoperative Chemotherapy, as Measured by the Total Number of Positive Nodes (SLN+ALND)
Description: Node status of patients after preoperative chemotherapy, as measured by the total number of positive nodes (SLN+ALND). Patients will be classified as node positive if they were determined to have at least one positive lymph node by SLN or ALND.
Time Frame: At time of surgery
Population: Patients with post-chemotherapy AUS results were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Post-chemotherapy AUS Suspicious: Patients with lymph nodes with abnormal morphology on AUS were classified as suspicious.
Arm/Group | Post-chemotherapy AUS Normal | Post-chemotherapy AUS Suspicious
Number analyzed (Participants) | 430 | 181
Participants
  0 | 171 | 47
  1-3 | 173 | 89
  4-10 | 42 | 28
  >10 | 10 | 7
  Missing/Unknown | 34 | 10
Statistical Analysis 1: Comparison: Post-chemotherapy AUS Normal vs Post-chemotherapy AUS Suspicious; Test type: Superiority; p = 0.003, t-test, 2 sided

5. Secondary Outcome: Pathologic Complete Nodal Response (pCR) Rate
Description: Pathologic complete nodal response (pCR) rate (percentage) wherein a nodal pCR is pathologically node-negative (pN0) on the basis of SLN surgery and ALND. A 95% binomial confidence interval was constructed for the pCR rate.
Time Frame: At the time of surgery
Population: Patients in cN1 and cN2 Cohort who had at least two SLNs excised and went on to complete ALND were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of SLN surgery/ALND
Arm/Group | cN1 Cohort | cN2 Cohort
Number analyzed (Participants) | 525 | 26
percentage of SLN surgery/ALND | 41.0 [36.7 to 45.3] | 46.1 [26.6 to 66.6]

6. Secondary Outcome: Residual Cancer Burden Class
Description: Residual cancer burden (RCB) is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. The calculated RCB index value can also be categorized as one of four RCB classes. The number of patients classified in the four RCB classes along with the number of patients missing this data by cohort are reported below. RCB of 0 represents a path complete response while increasing levels (I, then II, then III) indicate an increase in the 'amount' of residual disease remaining.
Time Frame: At time of surgery
Measure: Number; unit: participants
Arm/Group | cN1 Cohort | cN2 Cohort
Number analyzed (Participants) | 663 | 38
participants
  missing data | 162 | 6
  0 | 182 | 13
  I | 33 | 0
  II | 136 | 10
  III | 150 | 9

7. Other Pre Specified Outcome: Disease-Free Survival
Time Frame: Up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1-2 weeks post surgery
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation & scientific analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who started treatment & were evaluated for AEs. Serious AE (SAE) reports may include any secondary serious/non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and are in the SAE table.
Arm/Group | cN1 Cohort | cN2 Cohort
All-Cause Mortality (participants affected / at risk) | 1/676 | 0/39
Serious Adverse Events (participants affected / at risk) | 6/676 | 0/39
Other Adverse Events (participants affected / at risk) | 192/676 | 9/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cN1 Cohort (N=676) | cN2 Cohort (N=39)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cN1 Cohort (N=676) | cN2 Cohort (N=39)
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 (10) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (13) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (15) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 15 (15) | 0 (0)
Fatigue (General disorders) | 41 (41) | 3 (3)
Fever (General disorders) | 5 (5) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 54 (54) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 3 (3) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 6 (6) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 16 (16) | 2 (2)
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 19 (19) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (22) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 7 (7) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 46 (46) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 8 (8) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 39 (39) | 2 (2)
Ovulation pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Chest wall necrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 11 (11) | 0 (0)
Hot flashes (Vascular disorders) | 4 (4) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes